CLINICAL TRIAL: NCT02597660
Title: A Double-Blind Placebo-Controlled Study to Evaluate the Efficacy of Somatropin in the Treatment of Patellar Tendinopathy
Brief Title: A Study to Evaluate the Efficacy of Somatropin in the Treatment of Patellar Tendinopathy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI decided not to enroll
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: HUM00107019
Record Dates: First submitted 2015-11-03; First posted 2015-11-05 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2020-11

CONDITIONS: Tendinopathy
Keywords: patellar tendinopathy; somatropin; jumper's knee
MeSH Terms: conditions — Tendinopathy | interventions — Human Growth Hormone; Growth Hormone; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug: Somatropin (Active Comparator): Under ultrasound guidance, patients will receive an injection of somatropin (0.1mg in a volume of 0.2mL of bacteriostatic saline) into the area of tendinopathic lesion. A series of three injections will be delivered one week apart. Vials will be blinded.
  Interventions: Drug: Somatropin; Other: Progressive exercise program; Procedure: Patellar tendon biopsy
- Drug: Placebo (Placebo Comparator): Under ultrasound guidance, patients will receive an injection of 0.2mL of bacteriostatic saline (which is an equivalent volume of diluent used in the active comparator arm) into the area of tendinopathic lesion. A series of three injections will be delivered one week apart. Vials will be blinded.
  Interventions: Drug: Bacteriostatic saline; Other: Progressive exercise program; Procedure: Patellar tendon biopsy

INTERVENTIONS:
Drug: Somatropin — Active drug
  Other Names: Growth hormone; Human growth hormone
  Arms: Drug: Somatropin
Drug: Bacteriostatic saline — Placebo, the diluent used to reconstitute somatropin
  Other Names: Saline; 0.9% NaCl
  Arms: Drug: Placebo
Other: Progressive exercise program — Over a 12 week period beginning at the second study visit patients will perform a standard of care eccentric exercise training regime. Each session consists of three bilateral exercises: leg press, back squat, and hack squat. Subjects will complete four sets in each exercise with a 2-3 minute rest between sets. The repetitions/loads are: 15 repetition maximum (RM) week 1, 12RM weeks 2-3, 10RM weeks 4-5, 8RM weeks 6-8 and 6RM weeks 9-12. All exercises are performed from complete 0º to 90º of knee flexion and back again. Each of the eccentric and concentric phases will occur over a period of 3 seconds, respectively for a total of 6 seconds per contraction.
Procedure: Patellar tendon biopsy — Bilateral biopsies will be performed on an elective basis, although the investigators will aim to have 8 subjects in each group receive the biopsy. Biopsies will be obtained at the 26 week time point. The data obtained from the biopsy will help address the mechanism behind observed changes in outcome scores, physical measurements or imaging studies. The biopsy will be performed under ultrasound guidance and using sterile technique with a disposable 14G, 2cm biopsy instrument.

SUMMARY:
Patellar tendinopathy is one of the most frequent causes of non-traumatic knee pain and reduced function in patients. Standard treatment options for patellar tendinopathies include non-steroidal anti-inflammatory drugs, corticosteroids, cryotherapy, manual therapy, eccentric exercises, and ultrasound. Unfortunately many patients fail to respond to these therapies and return to normal activity levels, and recurrence rates for those who do respond are unacceptably high. Many patients who fail to respond display persistent degenerative changes on imaging studies suggesting a failure to regenerate the pathological tissue. Developing new therapies that can directly promote the synthesis of new, healthy extracellular matrix tissue could therefore address an important therapeutic need and make a substantial improvement in our ability to effectively treat patellar tendinopathy and reduce recurrence rates. Somatropin (human growth hormone of recombinant DNA origin) has been shown to increase protein synthesis and matrix production when delivered directly into the tendon. This study will evaluate the ability of somatropin to improve clinical outcomes and tissue quality in patients with chronic tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 18 - 50
* Patients with a greater than 3 month history of anterior knee pain
* Patients with a confirmed diagnosis of patellar tendinopathy (confirmation by ultrasonography demonstrating local anterior-posterior thickening of the tendon of at least 1mm compared with the mid-tendon level, and a hypo-echoic area)

Exclusion Criteria:

* Patients who have received corticosteroid injections within 12 months
* Patients who have full-width disruptions of the patellar tendon
* Patients who have undergone previous knee surgery or intraarticular injury
* Patients who have have arthritis (Kellgren and Lawrence grade 2 or higher), open growth plates, diabetes, cardiovascular disease, history of cancer or any major medical illnesses or endocrine disorders
* Patients with a body mass index greater than 35
* Women who are pregnant or planning to become pregnant
* Patients who are current collegiate, professional or elite athletes, or are participating in sports organizations that currently ban the use of somatropin

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Victorian Institute of Sport Assessment Patellar outcome score from enrollment | Week 1 to week 26

SECONDARY OUTCOMES:
Change in patient completed visual analog scale (VAS) of knee pain levels | Week 1, 2, 3, 4, 9, 14, 26
Change in patient completed Victorian Institute of Sport Assessment Patellar outcome score | Week 1, 2, 3, 4, 9, 14, 26
Change in patient completed Patient Reported Outcomes Measurement Instrument System (PROMIS) Physical Function Computer Adaptive Test | Week 1, 2, 3, 4, 9, 14, 26
Change in patient completed Patient Reported Outcomes Measurement Instrument System (PROMIS) Short Form Global Health Scale | Week 1, 2, 3, 4, 9, 14, 26
Ultrasound assessment of patellar tendon quality | Weeks 1, 14, 26
  Five point assessment scale of tendon quality (0 Normal, Normal tendon structure; 1 Mild, Ill-defined abnormal hypoechogenicity; 2 Moderate, Well-defined abnormal hypoechogenicity; 3 Severe, Well-defined abnormal hypoechogenicity and anechoic clefts; 4 Complete, Full-width tendon disruption or tear)
Electron micrographs of patellar tendon biopsy sample | Week 26
  Bilateral biopsies will be taken, and the size (measured in squared nanometers) will be measured
Gene expression of patellar tendon biopsy sample | Week 26
  Bilateral biopsies will be taken, and the expression of genes will be measured with microarrays or RNA-sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L Mendias, PhD, ATC, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Boesen AP, Dideriksen K, Couppe C, Magnusson SP, Schjerling P, Boesen M, Aagaard P, Kjaer M, Langberg H. Effect of growth hormone on aging connective tissue in muscle and tendon: gene expression, morphology, and function following immobilization and rehabilitation. J Appl Physiol (1985). 2014 Jan 15;116(2):192-203. doi: 10.1152/japplphysiol.01077.2013. Epub 2013 Nov 14. PMID 24235105
- [Background] Boesen AP, Dideriksen K, Couppe C, Magnusson SP, Schjerling P, Boesen M, Kjaer M, Langberg H. Tendon and skeletal muscle matrix gene expression and functional responses to immobilisation and rehabilitation in young males: effect of growth hormone administration. J Physiol. 2013 Dec 1;591(23):6039-52. doi: 10.1113/jphysiol.2013.261263. Epub 2013 Sep 30. PMID 24081158
- [Background] Gumucio JP, Sugg KB, Mendias CL. TGF-beta superfamily signaling in muscle and tendon adaptation to resistance exercise. Exerc Sport Sci Rev. 2015 Apr;43(2):93-9. doi: 10.1249/JES.0000000000000041. PMID 25607281
- [Background] Heinemeier KM, Mackey AL, Doessing S, Hansen M, Bayer ML, Nielsen RH, Herchenhan A, Malmgaard-Clausen NM, Kjaer M. GH/IGF-I axis and matrix adaptation of the musculotendinous tissue to exercise in humans. Scand J Med Sci Sports. 2012 Aug;22(4):e1-7. doi: 10.1111/j.1600-0838.2012.01459.x. Epub 2012 Mar 19. PMID 22429205
- [Background] Kongsgaard M, Kovanen V, Aagaard P, Doessing S, Hansen P, Laursen AH, Kaldau NC, Kjaer M, Magnusson SP. Corticosteroid injections, eccentric decline squat training and heavy slow resistance training in patellar tendinopathy. Scand J Med Sci Sports. 2009 Dec;19(6):790-802. doi: 10.1111/j.1600-0838.2009.00949.x. Epub 2009 May 28. PMID 19793213
- [Background] Visentini PJ, Khan KM, Cook JL, Kiss ZS, Harcourt PR, Wark JD. The VISA score: an index of severity of symptoms in patients with jumper's knee (patellar tendinosis). Victorian Institute of Sport Tendon Study Group. J Sci Med Sport. 1998 Jan;1(1):22-8. doi: 10.1016/s1440-2440(98)80005-4. PMID 9732118
- [Background] Hung M, Stuart AR, Higgins TF, Saltzman CL, Kubiak EN. Computerized Adaptive Testing Using the PROMIS Physical Function Item Bank Reduces Test Burden With Less Ceiling Effects Compared With the Short Musculoskeletal Function Assessment in Orthopaedic Trauma Patients. J Orthop Trauma. 2014 Aug;28(8):439-43. doi: 10.1097/BOT.0000000000000059. PMID 24378399
- [Derived] Lopes AD, Rizzo RR, Hespanhol L, Costa LO, Kamper SJ. Exercise for patellar tendinopathy. Cochrane Database Syst Rev. 2025 May 27;5(5):CD013078. doi: 10.1002/14651858.CD013078.pub2. PMID 40421598